CLINICAL TRIAL: NCT02571036
Title: A Multicenter Phase 1, Open-Label Study of DCC-2618 to Assess Safety, Tolerability, Efficacy, and Pharmacokinetics in Patients With Advanced Malignancies
Brief Title: A Safety, Tolerability and PK Study of DCC-2618 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2618-01-001
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Gastrointestinal Stromal Tumors; Advanced Systemic Mastocytosis; Advanced Cancers
Keywords: Gastrointestinal stromal tumors (GIST); systemic mastocytosis (SM); PDGFR-alpha; KIT; mast cell leukemia (MCL); mast cell disease (MCD); DCC-2618; melanoma; aggressive systemic mastocytosis (ASM); soft tissue sarcoma (STS); germ cell tumors; penile cancer; non-small cell lung carcinoma (NSCLC); renal impairment; malignant gliomas
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Mastocytosis, Systemic; Leukemia, Mast-Cell; Mast Cell Activation Disorders; Melanoma; Sarcoma; Neoplasms, Germ Cell and Embryonal; Penile Neoplasms; Carcinoma, Non-Small-Cell Lung; Renal Insufficiency; Glioma | interventions — ripretinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (12):
- Escalation (Experimental): Escalation Phase: DCC-2618 tablets in escalating dose cohorts given orally BID (twice daily) every 12 hours or once daily (QD) for repeated 28-day cycles. Participants may continue to receive study drug until discontinuation criteria are met. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 1 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with GIST who have received 3 prior therapies. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 2 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with GIST who have received 4 prior therapies. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 3 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with GIST who have received at least one prior therapy and no more than 2 prior therapies. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 4 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with systemic mastocytosis and other hematologic malignancies.[Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 5 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with malignant gliomas.[Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 6 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with other solid tumors. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 7 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with melanomas. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 8 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with soft tissue sarcomas.[Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 9 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with germ cell, penile cancer and non-small cell lung carcinoma (NSCLC). [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Expansion Cohort 10 (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles in patients with GIST and other solid tumors with renal impairment. [Closed for Enrollment]
  Interventions: Drug: DCC-2618
- Extension Cohort (Experimental): 150 mg DCC-2618 given once daily in repeated 28-day cycles for active patients from the Escalation and Extension Phases.
  Interventions: Drug: DCC-2618

INTERVENTIONS:
Drug: DCC-2618 — 50 mg formulated tablets
  Other Names: ripretinib
  Arms: Expansion Cohort 1; Expansion Cohort 10; Expansion Cohort 2; Expansion Cohort 3; Expansion Cohort 4; Expansion Cohort 5; Expansion Cohort 6; Expansion Cohort 7; Expansion Cohort 8; Expansion Cohort 9; Extension Cohort
Drug: DCC-2618 — 10 mg and 50 mg formulated tablets
  Other Names: ripretinib
  Arms: Escalation

SUMMARY:
This is a Phase 1, open-label, first-in-human (FIH) dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of DCC-2618, administered orally (PO), in adult patients with advanced malignancies. The study consists of 2 parts, a dose-escalation phase, and an expansion phase. All active patients (from both dose-escalation and expansion phases) will then transition into an extension phase.

ELIGIBILITY:
Inclusion Criteria (Escalation and Expansion Phases)

Patients must meet the following criteria to be eligible to enroll in the study:

1. Male or female patients ≥18 years of age.
2. Patients must have histologically confirmed solid tumors or hematologic malignancies. Eligible patients include the following:

   1. GIST patients must have a KIT and PDGFRA mutation and must have progressed on or had an intolerability to at least 1 line of systemic anticancer therapy.
   2. SM patients must have a confirmed diagnosis of advanced SM according to 2016 World Health Organization (WHO) criteria for SM and must have documented KIT mutant disease. Patients with imatinib-sensitive KIT mutations must have progressed on or were intolerant to a tyrosine kinase inhibitor. Patients with advanced SM must present with at least 1 eligible C-Finding (organ damage) per 2013 International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) & European Competence Network on Mastocytosis consensus response criteria; please see below for MCL exception.

   Advanced SM includes:

   i. Aggressive SM (ASM)

   ii. SM with associated hematologic neoplasm (SM-AHN), wherein the AHN does not require immediate alternative therapy. AHNs that are eligible include: low grade myelodysplastic syndrome (MDS) with a high SM burden who require treatment for SM only, myeloproliferative neoplasms (MPN), MDS/MPN, unclassifiable MDS, and HES/CEL.

   iii. MCL

   • Patients with histopathologically-confirmed MCL without a C-finding are eligible.

   iv. Symptomatic SSM

   • By definition, SSM patients must have at least 2 B-findings, and clinically significant symptom burden (eg, flushing, diarrhea, etc.) despite maximal treatment with approved agents to treat mediator symptoms, such as antihistamines and cromolyn sodium.

   v. Patients with hematologic malignancies featuring clonal expansion of eosinophils driven by genomic alterations of KIT or PDGFRA (eg, HES or CEL) are eligible if they have progressed on or are intolerant of imatinib therapy. Patients with de novo imatinib resistant mutations, such as but not limited to KIT D816V or PDGFRA D842V, are eligible without prior imatinib therapy.

   c. Malignant glioma patients with genomic alterations potentially conferring sensitivity to DCC-2618 including, but not limited to, amplification and/or mutations of PDGFRA and/or KIT.

   Other solid tumor patients that have alterations in genes encoding kinases that are targets of DCC-2618. This includes:
   * Melanoma
   * Soft tissue sarcoma patients (including but not limited to: malignant peripheral nerve sheath tumors (MPNST), desmoplastic small round cell tumors (DSRCT), and dermatofibrosarcoma protuberans tumors (DFSP)
   * Other solid tumor patients (non-melanoma, non-STS; specifically germ-cell, penile, and non-small cell lung carcinoma)
   * Renal impairment cohort
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2.
4. Adequate organ function and bone marrow function.

Exclusion Criteria (Escalation and Expansion Phases)

Patients meeting any of the following criteria will be excluded from the study:

1. GIST patients with wild type or unknown KIT or PDGFRA status.
2. Patients with SM or other hematologic malignancies will be excluded if the following apply:

   1. SM patients with neutropenia accompanied by fever or infection, or thrombocytopenia associated with clinically significant bleeding.

      • Patients with an infection that is well controlled with antibiotics are eligible if there is an immediate need for treatment.
   2. SM-AHN patients diagnosed with:

   i. SM with MDS who require treatment for MDS. ii. Patients requiring immediate treatment for AHN.

   c. Patients with leukemias, with the exception of MCL and CEL, that have progressed after imatinib.

   d. Eosinophilic myeloproliferative neoplasm patients: i. Lacking a mutation that is a known target of DCC-2618.
3. Prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of DCC-2618. Patients receiving adjuvant cancer treatment are not eligible if those medications are potentially active against GIST or excluded per protocol.
4. New York Heart Association class III and IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure.
5. Arterial thrombotic or embolic events such as cerebrovascular accident (including ischemic attacks) or hemoptysis within 6 months before start of study drug.
6. Venous thrombotic events (eg, deep vein thrombosis) or pulmonary arterial events (eg, pulmonary embolism) within the 3 months before start of study drug. Patients with venous thrombotic events ≥3 months before start of study drug on stable anticoagulation therapy are eligible.
7. Baseline prolongation of the rate-corrected QT interval based on repeated demonstration of QT interval corrected by Fridericia's formula (QTcF) >450 ms in males or >470 ms in females or history of long QT interval corrected (QTc) syndrome.
8. Left ventricular ejection fraction (LVEF) <50% or below the lower limit of normal (whichever is higher).
9. Major surgery within 4 weeks of the first dose of study drug; following major surgeries >4 weeks prior to the first dose of study drug, all surgical wounds must be healed and free of infection or dehiscence.
10. Any other clinically significant comorbidities.
11. Illnesses that could affect oral absorption.
12. Known human immunodeficiency virus or active hepatitis C infection only if the patient is taking per protocol prohibited medications, active hepatitis B, or active hepatitis C infection.
13. If female, the patient is pregnant or lactating.
14. Known allergy or hypersensitivity to any component of the investigational drug product. Patients with history of Stevens-Johnson syndrome on a prior tyrosine kinase inhibitor (TKI) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of oral DCC-2618: incidence of adverse events | Approximately 24 months
  Dose limiting toxicities, AEs, SAEs, discontinuation of drug due to toxicity, physical exams and ECOG PS, ophthalmologic examinations, changes from baseline in laboratory parameters, electrocardiograms, LVEF, and vital signs.
Determination of the Maximum Tolerated Dose and the Recommended Phase 2 Dose | 18 months
Expansion Phase: Assess Antitumor Activity of DCC-2618 in all diseases | Approximately 24 months
  Objective response rate (ORR); Disease control rate (DCR)

SECONDARY OUTCOMES:
Determine the PK profile of oral DCC-2618 | Predose and up to 24 hours postdose (Cycle = 28 Days)
Escalation Phase: Assess Antitumor Activity of DCC-2618 in patients with advanced malignancies | Approximately 24 months
  Objective response rate (ORR); Disease control rate (DCR)

CONTACTS AND LOCATIONS:
Overall Officials: Deciphera Pharmaceuticals, LLC, Study Director — Deciphera Pharmaceuticals, LLC
Locations (26):
- United States (16):
  - Honor Health (GIST, mastocytosis, other solid tumors), Scottsdale, Arizona
  - UCLA Hematology Center (mastocytosis), Los Angeles, California
  - UCLA (glial malignancies only), Los Angeles, California
  - Stanford University Comprehensive Cancer Center (GIST), Palo Alto, California
  - Stanford University Hematology Clinic (mastocytosis), Palo Alto, California
  - UCSF (glial malignancies only), San Francisco, California
  - Mayo Clinic (GIST, mastocytosis, glial malignancies, other solid tumors), Jacksonville, Florida
  - University of Miami (GIST, mastocytosis, glial malignancies, other solid tumors), Miami, Florida
  - Dana Farber Cancer Institute (GIST, mastocytosis, glial malignancies, other solid tumors), Boston, Massachusetts
  - Colombia University Medical Center (mastocytosis), New York, New York
  - Memorial Sloan Kettering Cancer Center (GIST, mastocytosis, glial malignancies, other solid tumors), New York, New York
  - OHSU (GIST & mastocytosis only), Portland, Oregon
  - Fox Chase Cancer Center (GIST only), Philadelphia, Pennsylvania
  - MD Anderson Cancer Center (GIST, mastocytosis, glial malignancies, other solid tumors), Houston, Texas
  - Huntsman Cancer Institute (GIST, mastocytosis, glial malignancies, other solid tumors), Salt Lake City, Utah
  - Virginia Commonwealth University School of Medicine (mastocytosis), Richmond, Virginia
- Princess Margaret Cancer Centre (GIST, other solid tumors), Toronto, Canada
- Germany (5):
  - Uniklinik RWTH Aachen (mastocytosis, GIST, and other solid tumors), Aachen
  - HELIOS Klinikum Berlin-Buch (GIST, and other solid tumors), Berlin
  - Essen University Hospital (mastocytosis, GIST, and other solid tumors), Essen
  - Freiburg University Hospital (mastocytosis, and other solid tumors), Freiburg im Breisgau
  - University Medical Centre Mannheim (mastocytosis), Mannheim
- University Hospital of Verona (mastocytosis), Verona, Italy
- Leiden University Medical Center (GIST and other solid tumors), Leiden, Netherlands
- United Kingdom (2):
  - Guy's Hospital (mastocytosis only), London
  - Royal Marsden Hospital (GIST, glial malignancies, other solid tumors), London

REFERENCES:
- [Derived] Janku F, Abdul Razak AR, Chi P, Heinrich MC, von Mehren M, Jones RL, Ganjoo K, Trent J, Gelderblom H, Somaiah N, Hu S, Rosen O, Su Y, Ruiz-Soto R, Gordon M, George S. Switch Control Inhibition of KIT and PDGFRA in Patients With Advanced Gastrointestinal Stromal Tumor: A Phase I Study of Ripretinib. J Clin Oncol. 2020 Oct 1;38(28):3294-3303. doi: 10.1200/JCO.20.00522. Epub 2020 Aug 17. PMID 32804590